CLINICAL TRIAL: NCT05659732
Title: A Phase 1b Study of PEP07 (Checkpoint Kinase 1 Inhibitor) in Patients With Advanced Cancer
Brief Title: A Study of PEP07 (Checkpoint Kinase 1 Inhibitor) in Patients With Advanced Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: PharmaEngine (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PEP07-101
Record Dates: First submitted 2022-11-30; First posted 2022-12-21 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Acute Myeloid Leukemia; Lymphoma, Mantle-Cell
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Lymphoma, Mantle-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PEP07 Monotherapy (Arm A) (Experimental): The dose finding of PEP07 monotherapy consists of an accelerated dose escalation followed by a standard "3+3" dose escalation. Accelerated titration will continue until 1 patient experiences a DLT, or ≥ grade 2 AE related to PEP07 (except for hematologic toxicities) at any dose level, after which, additional 2 patients will be enrolled in the same cohort, and the study will be switched to a 3+3 scheme.
  Expansion cohorts with 12 patients will be opened for Arm A at the RP2D once efficacy signal is observed at this level.
  Interventions: Drug: PEP07

INTERVENTIONS:
Drug: PEP07 — PEP07 is a selective Chk1 inhibitor maleate drug which is supplied as a hard gelatin capsule. PEP07 will be provided as 20 mg and 150 mg strength capsules to be administrated orally. Patients allocated to different dose levels of PEP07 monotherapy will receive either 20 mg or 150 mg oral capsules for 2 consecutive days followed by 5 days treatment off (2-on/5-off) schedule every week, 4 weeks as a treatment cycle.

SUMMARY:
The goal of this clinical trial is

* To assess the safety and tolerability of PEP07 administered orally as a single dose and at escalating dose levels, and, to determine the dose-limiting toxicity (DLT) of study treatment in patients with Acute Myeloid Leukemia (AML) and Mantle Cell Lymphoma (MCL).
* To determine the maximum tolerated dose (MTD) and/or recommended Phase 2 dose (RP2D) of PEP07 monotherapy.

Participants will receive PEP07 administered orally once daily (QD) for 2 consecutive days and 5 days off, every week for 4 weeks until disease progression, intolerable toxicity, confirmed pregnancy, death, consent withdrawal, HSCT or other anti-cancer treatment is required, or the Sponsor ends the study, whichever occurs first.

DETAILED DESCRIPTION:
This is a Phase 1b, open-label, multi-center study recruiting patients with R/R AML and MCL.

The study will utilize an Accelerated Titration Design in the lower dose levels followed by a traditional 3+3 dose escalation design at higher dose levels until RP2D is determined. The starting dose will be 40 mg.

All potential study candidates will provide informed consent and will undergo screening procedures before participating in the study. After a screening period of up to 28 days, qualified patients will be enrolled to receive their assigned dose regimen of PEP07 monotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Must be ≥ 18 years of age.
2. Must have histological or cytological confirmation advanced hematologic malignancy including:

   * Relapsed or refractory AML (by the 5th edition of World Health Organization [WHO] classification of Hematolymphoid tumors)
   * OR Relapsed or refractory MCL and have received at least two prior lines of treatment, including chemoimmunotherapy and BTKi and at least 1 measurable site of disease according to Revised Response Criteria for Malignant Lymphoma.
3. Must have Eastern Cooperative Oncology Group (ECOG) Performance score of 0 to 2.
4. Must have adequate renal function as demonstrated by a calculated creatinine clearance ≥ 50 mL/min; determined via urine collection for 24-hour creatinine clearance or by the Cockcroft Gault formula.
5. Must have adequate liver function as demonstrated by:

   * aspartate aminotransferase (AST) ≤ 2.5 × ULN
   * alanine aminotransferase (ALT) ≤ 2.5 × ULN
   * bilirubin ≤ 1.5 × ULN (unless considered due to leukemic organ involvement. Patients with Gilbert's Syndrome may have had a bilirubin > 1.5 × ULN per discussion between the PI or designee and sponsor)
6. Left ventricular ejection fraction (LVEF) ≥ 50% measured by multiple-gated acquisition (MUGA) or echocardiogram.
7. Previous AEs have been improved to baseline or Grade ≤ 1 NCI CTCAE v5.0.
8. Female patients with reproductive potential must have a negative serum pregnancy test 7 days prior to the administration of PEP07.
9. Patients will be required to have a Covid negative test either via reverse transcriptase polymerase chain reaction (RTPCR) or a rapid antigen test (RAT) test on Day -7/Day 1.
10. Provision of signed and dated informed consent form.

Exclusion Criteria:

1. Pregnant or breastfeeding females
2. Females of childbearing potential and males whose partners are of childbearing potential who do not agree to the use of 2 forms of highly effective contraception during the treatment period and for 120 days after the last dose of PEP07.
3. Patients who have received anti-cancer therapy including chemotherapy, radiotherapy, hormonal, or any investigational therapy within 14 days or 5 half-lives (whichever is shorter), or immunotherapy within 30 days prior to the first dose of PEP07. Patients who have received hydroxyurea or dexamethasone at any time prior to the start of study treatment is an exception to this criterion.
4. Patients who have undergone allogeneic hematopoietic stem cell transplant (HSCT) within 60 days of PEP07 treatment.
5. Patients who have received strong or moderate CYP3A4 inhibitors or inducers such as ketoconazole, erythromycin, netupitant, isavuconazole etc. within 5 half-lives or 7 days (whichever is the shortest) prior to the initiation of study treatment.
6. Viral infection with HIV or viral hepatitis type B or C which require antiviral therapy and/or have positive serology test of hepatitis B surface antigen [HBsAg (+)] with HBV DNA ≥ 1000 IU/mL, or hepatitis C virus antibody [anti-HCV Ab (+)] with HCV RNA (+). If a patient is HBsAg (+) then HBV DNA needs to be tested. If a patient is anti-HCV Ab (+) then the patient needs to be followed for HCV RNA (-) to be enrolled.
7. Uncontrolled systemic infection /or requiring isolation.
8. Patients with previous history of other malignant diseases within the last 5 years (other than adequately treated non-melanotic skin cancer, in-situ carcinoma of the uterine cervix or myelodysplastic syndromes).
9. Patients with ongoing ≥ Grade 2 (CTCAE v5.0) toxicity (except alopecia and hot flashes) related to previous treatment.
10. Patients with baseline QTc interval > 450 msec (i.e., CTCAE Grade ≥ 2) at screening (within 28 days prior to 1st dose of PEP07, mean of triplicate readings within approximately 5 minutes).
11. Patients with cardiovascular disability status of New York Heart Association (NYHA) ≥ Class III, left ventricular ejection fraction < 45 % at baseline, history of cardiac ischemia within the past 6 months, or prior history of cardiac arrhythmia requiring treatment.
12. Patients who have undergone any major surgery within 3 weeks prior to first study drug administration after enrollment.
13. Patients with known active central nervous system (CNS) or leptomeningeal involvement.
14. Patients who have had any of the following within 6 months prior to first administration of PEP07 after enrollment: myocardial infarction, severe/unstable angina pectoris, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident or transient ischemic attack, or seizure disorder.
15. Have a history of hypersensitivity reactions or allergic reactions to PEP07 excipients and components.
16. Patients with other medical or psychiatric condition that, in the opinion of the investigator, might interfere with the patient's participation in the trial or interfere with the interpretation of trial results.
17. Others who are ineligible to participate in this clinical study as determined by the PI or designee.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2023-07-17 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
To assess the safety and tolerability of PEP07 administered orally as a single dose and at escalating dose levels, and, to determine the dose-limiting toxicity (DLT) of study treatment in patients with AML and MCL. | 4 weeks after first dosing
  to find out the DLT
To determine the maximum tolerated dose (MTD) and/or recommended Phase 2 dose (RP2D) of PEP07 monotherapy. | 4 weeks after first dosing
  to find out the MTD

SECONDARY OUTCOMES:
To assess the AUC from time zero to infinity (AUC0-inf) of single and multiple oral PEP07 as a monotherapy. | 6 months
  to know the PK profile
To assess the Time to maximum (peak) plasma concentration (Tmax) of single and multiple oral PEP07 as a monotherapy. | 6 months
  to know the PK profile
To assess the apparent half-life (t1/2) of single and multiple oral PEP07 as a monotherapy. | 6 months
  to know the PK profile
To assess the Maximum observed concentration (Cmax) of single and multiple oral PEP07 as a monotherapy. | 6 months
  to know the PK profile
To assess preliminary evidence of anti-tumor activity of PEP07 by progression free survival (PFS). | after first dosing to disease progression
  to know the efficacy
To assess preliminary evidence of anti-tumor activity of PEP07 by progression free survival (PFS). | after first dosing to disease progress
  to know the efficacy

OTHER OUTCOMES:
To assess Chk1 level in patients with AML and MCL. | 6 months
  to find out the the changes in biomarkers
To assess γH2AX level in patients with AML and MCL. | 6 months
  to find out the the changes in biomarkers
To assess pCHK1 level in patients with AML and MCL. | 6 months
  to find out the the changes in biomarkers

CONTACTS AND LOCATIONS:
Overall Officials: Hsin-An Hou, M.D., Principal Investigator — Division of Hematology, Department of Internal Medicine, National Taiwan University Hospital
Locations (5):
- Monash Medical Centre, Clayton, Victoria, Australia
- Taiwan (4):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - Chang Gung Memorial Hospital- Linkou, Taipei
  - National Taiwan University Hospital, Taipei